CLINICAL TRIAL: NCT05530473
Title: Combined Capsular Tension Ring and IOL Implantation for Management of Cataracts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Jin Yang, Professor, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOL&CTR
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Intraocular Lens Rotation; Capsular Tension Ring

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTR Group (Experimental): Eyes had a capsular tension ring (CTR) implanted into the capsular bag during the cataract surgery.
  Interventions: Device: capsular tension ring
- NCTR Group (No Intervention): Eyes underwent cataract surgery without implanting a CTR.

INTERVENTIONS:
Device: capsular tension ring — To insert a capsular tension ring during the cataract surgery
  Other Names: capsular tension ring (ACPi-11; Bausch&Lomb)
  Arms: CTR Group

SUMMARY:
This study included cataract patients who underwent intraocular lens (IOL) implantation with or without capsular tension ring (CTR), which aimed to evaluate the contribution of the use of CTR in clinical visual outcomes and rotational stability of IOL after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

-cataract

Exclusion Criteria:

* preexisting corneal pathology
* small pupil
* glaucoma
* zonular dehiscence
* a history of ocular trauma or surgery
* uveitis
* intraoperative complications

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
IOL rotation degree at one hour | one hour
  After the pupil was dilated, the IOL axis was recorded by a senior surgeon (C. L.) using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at 1 day | one day
  After the pupil was dilated, the IOL axis was recorded by a senior surgeon (C. L.) using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at 3 days | three days
  After the pupil was dilated, the IOL axis was recorded by a senior surgeon (C. L.) using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at 1 week | one week
  After the pupil was dilated, the IOL axis was recorded by a senior surgeon (C. L.) using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at 2 weeks | two weeks
  After the pupil was dilated, the IOL axis was recorded by a senior surgeon (C. L.) using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at 1 month | one month
  After the pupil was dilated, the IOL axis was recorded by a senior surgeon (C. L.) using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at 3 months | three months
  After the pupil was dilated, the IOL axis was recorded by a senior surgeon (C. L.) using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at 6 months | three months
  After the pupil was dilated, the IOL axis was recorded by a senior surgeon (C. L.) using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at 12 months | three months
  After the pupil was dilated, the IOL axis was recorded by a senior surgeon (C. L.) using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
Residual astigmatism (RAS) at two weeks | two weeks
  RAS after surgery, which was measured as manifest refraction at two weeks
Residual astigmatism (RAS) at one month | one month
  RAS after surgery, which was measured as manifest refraction at one month

SECONDARY OUTCOMES:
visual acuity (VA) at 1 day | two weeks
  Uncorrected distance visual acuity (UDVA) of participants after surgery at two weeks
visual acuity (VA) at 3 days | two weeks
  Uncorrected distance visual acuity (UDVA) of participants after surgery at two weeks
visual acuity (VA) at 1 weeks | two weeks
  Uncorrected distance visual acuity (UDVA) of participants after surgery at two weeks
visual acuity (VA) at 2 weeks | two weeks
  Uncorrected distance visual acuity (UDVA) of participants after surgery at two weeks
visual acuity (VA) at 1 month | one month
  Uncorrected distance visual acuity (UDVA) of participants after surgery at one month
visual acuity (VA) at 3 months | three months
  Uncorrected distance visual acuity (UDVA) of participants after surgery at three months
visual acuity (VA) at 6 months | six months
  Uncorrected distance visual acuity (UDVA) of participants after surgery at six months
visual acuity (VA) at 12 months | twelve months
  Uncorrected distance visual acuity (UDVA) of participants after surgery at twelve months
IOL tilt at 1 day | one day
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.
IOL tilt at 3 days | three days
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.
IOL tilt at 1 week | one week
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.
IOL tilt at 2 weeks | two weeks
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.
IOL tilt at 1 month | one month
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.
IOL tilt at 3 months | three months
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.
IOL tilt at 6 months | six months
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, PhD, Principal Investigator — Eye & ENT Hospital
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin X, Ma D, Han X, Hua Z, Shen W, Qiu X, Cai L, Yang J. Rotational stability of plate-haptic toric intraocular lenses implantation with a capsular tension ring: prospective randomized paired-eye study. J Cataract Refract Surg. 2025 Jan 1;51(1):31-39. doi: 10.1097/j.jcrs.0000000000001554. PMID 39353092